CLINICAL TRIAL: NCT06115265
Title: Ketogenic Diet and Diabetes Demonstration Project
Acronym: KDDP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Kristen M Gonzales, Assistant Professor, University of New Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-364
Record Dates: First submitted 2023-10-17; First posted 2023-11-02 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes; PreDiabetes; Obesity; Ketogenic Dieting
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Obesity | interventions — Diet, Ketogenic; Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: Subjects will be recruited to participate in either KDDP or NDPP. The lifestyle interventions are identical with the exception of dietary recommendations. Groups will be matched according to age, sex, and HbA1c.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KDDP (Experimental): KDDP - Participants enrolled in the KDDP arm will be placed on a traditional ketogenic diet (<20 grams of carbohydrate/day).
  Interventions: Behavioral: Ketogenic diet
- NDPP (Experimental): NDPP - Participants enrolled in the NDPP arm will be placed on a low fat diet.
  Interventions: Behavioral: Low Fat diet

INTERVENTIONS:
Behavioral: Ketogenic diet — KDDP and NDPP will deliver identical comprehensive lifestyle counseling and follow up to participants, but dietary interventions in each group will differ, with KDDP participants receiving a ketogenic diet and NDPP participants receiving a low fat diet.
  Arms: KDDP
Behavioral: Low Fat diet — KDDP and NDPP will deliver identical comprehensive lifestyle counseling and follow up to participants, but dietary interventions in each group will differ, with KDDP participants receiving a ketogenic diet and NDPP participants receiving a low fat diet.
  Arms: NDPP

SUMMARY:
KDDP is a prospective, 12-month pilot study comparing the effects of a novel lifestyle program, the Ketogenic Diet and Diabetes Demonstration Project (KDDP) to those of the National Diabetes Prevention Program (NDDP). KDDP is modeled to mimic the delivery platform of NDPP with the exception that participants in KDDP will be placed on a medically-supervised ketogenic diet, and participants in NDPP will be placed on a low fat diet.

The purpose of this study is to compare the metabolic effects of the KDDP and the NDPP on glycemic control, lipid parameters, blood pressure, heart rate, weight, and coronary artery calcium scores in individuals with either type 2 diabetes or prediabetes.

DETAILED DESCRIPTION:
KDDP is a prospective, 12-month pilot study comparing the effects of the KDDP vs. CDC NDPP in patients with obesity and dysglycemia. KDDP is the Ketogenic Diet and Diabetes Demonstration Project arm. Individuals enrolled in the KDDP arm will attend a mandatory Weight Management class through the Center for Diabetes and Nutrition Education, and they will participate in a standard comprehensive lifestyle intervention program that is identical to that of the NDPP with the exception of dietary recommendations. Individuals in the KDDP arm will be educated on and follow a ketogenic diet (<20g carbohydrates/day). They will receive guidance on tracking carbohydrate intake daily, and home point-of-care ketone breath testing will be performed at regular intervals to ensure that ketosis is being achieved and maintained. They will attend weekly educational sessions facilitated by trained dieticians. Individuals enrolled in the CDC NDPP arm will adhere to a low fat diet and receive identical follow up with the dieticians relative to those enrolled in the KDDP arm. Individuals in both arms will be matched for age, sex, weight, and A1c.

Baseline measures at study entry will include weight, height, systolic and diastolic blood pressure, heart rate, hemoglobin A1c, fasting plasma glucose, total cholesterol, triglycerides, HDL cholesterol, and LDL cholesterol. These parameters will be measured every 3 months throughout the study and at study completion. Additionally, participants in both groups will be consented to undergo CAC scanning at baseline and at 12 months to assess for any differences in dietary interventions on CAC scores.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years old
* BMI ≥27 kg/m2
* Hemoglobin A1c ≥ 5.7% and/or fasting plasma glucose of 100-125 mg/dL

Exclusion Criteria:

* Known clinical cardiovascular disease (i.e. prior stroke, myocardial infarction, peripheral artery disease)
* LDL cholesterol ≥ 190 mg/dL
* Triglycerides ≥ 500 mg/dL
* History of type 1 diabetes
* History of diabetic ketoacidosis
* Individuals requiring insulin
* Advanced renal disease
* Advanced liver disease
* Terminal cancer
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Weight in kg | 12 months
  Change in weight over 12-months in KDDP arm vs NDPP arm

SECONDARY OUTCOMES:
Blood pressure in mmHg | 12 months
  Changes in the above measures from baseline to 12 months in KDDP arm vs. NDPP arm
Heart rate in beats per minute (BPM) | 12 months
  Changes in heart rate from baseline to 12 months in KDDP arm vs. NDPP arm
HbA1c as a percent | 12 months
  Changes in HbA1c from baseline to 12 months in KDDP arm vs. NDPP arm
Fasting lipids in mg/dL | 12 months
  Changes in fasting lipids from baseline to 12 months in KDDP arm vs. NDPP arm
Fasting plasma glucose in mg/dL | 12 months
  Changes in fasting plasma glucose from baseline to 12 months in KDDP arm vs. NDPP arm
CAC scores | 12 months
  Changes in CAC scores from baseline to 12 months in KDDP arm vs. NDPP arm

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Gonzales, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared with researchers outside of those directly conducting this study.